CLINICAL TRIAL: NCT00989599
Title: Therapeutic Topic Use of Chamomilla Recutita in Phlebitis Due to Peripheral Intravenous Therapy
Brief Title: Use of Chamomilla Recutita in Phlebitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Paula Elaine Diniz dos Reis, Escola de Enfermagem de Ribeirão Preto - USP
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: USPRecutita-01
Record Dates: First submitted 2009-10-02; First posted 2009-10-05 (Estimated); Last update posted 2009-10-05 (Estimated); Status verified 2009-10

CONDITIONS: Phlebitis
Keywords: phlebitis; Chamomilla recutita; Catheterization peripheral
MeSH Terms: conditions — Phlebitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- compress of Chamomilla recutita infusion (Experimental): Patients who developed phlebitis due to peripheral intravenous infusion in anti-neoplasm chemotherapy were treated with a compress of Chamomilla recutita infusion for 20 minutes three times per day
  Interventions: Other: compress of Chamomilla recutita infusion
- compress of lukewarm water (Active Comparator): Patients with phlebitis due to peripheral intravenous infusion in anti-neoplasm chemotherapy, in control group, were treated with a compress of lukewarm water for 20 minutes three times per day
  Interventions: Other: compress of lukewarm water

INTERVENTIONS:
Other: compress of Chamomilla recutita infusion — Patients with phlebitis due to peripheral intravenous infusion in anti-neoplasm chemotherapy were treated with a compress of Chamomilla recutita infusion for 20 minutes three times per day
  Arms: compress of Chamomilla recutita infusion
Other: compress of lukewarm water — Patients with phlebitis due to peripheral intravenous infusion in anti-neoplasm chemotherapy, in control group, were treated with a compress of lukewarm water for 20 minutes three times per day
  Arms: compress of lukewarm water

SUMMARY:
To verify the efficacy of topical applications of Chamomilla recutita infusion for phlebitis treatment, before dose response curve study and pilot study.

DETAILED DESCRIPTION:
The hypothesis adopted was that patients with phlebitis due to peripheral intravenous infusion in anti-neoplasm chemotherapy, treated with a compress of Chamomilla recutita infusion for 20 minutes three times per day, would present a shorter phlebitis regression time in comparison with patients treated with a lukewarm water compress.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with cancer who had infusion phlebitis during the administration of intravenous chemotherapy peripheral under hospitalization.

Exclusion Criteria:

* Report made by the subject of study, prior hypersensitivity reaction or presentation during the research, adverse reaction to chamomile or any plant of the family Asteraceae ou Compositae: margarida (Aster tripolium), crisântemo (Chrysanthemum leucanthemum), artemísia or isopo santo (Artemísia vulgaris), carpineira or ambrósia americana (Ambrosia artemisiifolia) and senécio (Senecio jacobaea L.);
* Prescription during the process of data collection, some kind of anti-inflammatory with systemic or topical activity where it was located phlebitis, and, upon the occurrence of bacterial phlebitis, had been prescribed topical or systemic antibiotic therapy;
* Refusal of the subject to participate in the study, regardless of the time.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2004-09; Primary Completion 2007-12 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
phlebitis regression time | medium of 7 days

SECONDARY OUTCOMES:
palpable venous cord regression time | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Paula ED Reis, RN, PhD, Principal Investigator — University of Sao Paulo; Emília C Carvalho, RN, MsC, PhD, Study Director — University of Sao Paulo
Locations (1):
- Hospital de Base do Distrito Federal, Brasília, Brasília/DF, Brazil